CLINICAL TRIAL: NCT06073691
Title: Intermittent Anaerobic Exercise as Interoceptive Exposure Strategy in the Treatment of Patients With Panic Disorder: Randomized Clinical Trial
Brief Title: Interoceptive Exposure in Panic Disorder
Acronym: IEPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IPq-HCFMUSP
Record Dates: First submitted 2023-09-20; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-09

CONDITIONS: Panic Attacks and Disorders
Keywords: aerobic exercise; physical activity; treatment; interoception; exposure therapy.
MeSH Terms: conditions — Panic Disorder; Disease; Motor Activity

STUDY DESIGN:
Intervention Model Description: The study was designed as a prospective, two-arms, blinded, randomized controlled clinical trial. Patients and evaluators were informed that the participants might receive an active pharmacological treatment or a matching placebo; however, all patients received only a placebo. The study was conducted at the Anxiety Disorder Program of the Institute of Psychiatry and at the Institute of Orthopaedics and Traumatology of the University of Sao Paulo Medical School, Sao Paulo, Brazil.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise intervention (Experimental): On each training day, the activity started with a 5-minute stretching and warm-up session; then, a 15-minute walk at 65% of the maximum heart rate (MHR), followed by a 30-second run at 85% MHR, and finally another 15-minute walk at 65% MHR. The running time was gradually increased in individualized and supervised sessions. The exercise intensity was predetermined based on the patient's baseline cardiopulmonary function, and the heart rates (HR) were assessed using a Polar RS300X heart rate monitor.
  Interventions: Behavioral: Exercise intervention
- Placebo (Placebo Comparator): The participants might receive an active pharmacological treatment or a matching placebo
  Interventions: Behavioral: Exercise intervention; Other: Placebo

INTERVENTIONS:
Behavioral: Exercise intervention — Practice systematic and regular aerobic physical exercise (walking and running).
  Other Names: Interoceptive exposure therapy
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to test action exercises in the treatment of people with a diagnosis of Panic disorders with or without agoraphobia.

The main question it aims to answer is:

To investigate the feasibility and effectiveness of a Panic Disorder (PD) treatment protocol based on anaerobic exercise as an interoceptive exposure therapy.

Participants will The participants were randomly allocated to a 12-week program of either Intermittent Anaerobic Exercise.

Researchers will compare two groups, one with treatment through an intermittent aerobic exercise (IAE) protocol and the other group with treatment via a muscle relaxation protocol (RT), to see if there is feasibility and efficacy of a Panic Disorder treatment protocol based on anaerobic exercise as exposure therapy, compared to a relaxation activity.

DETAILED DESCRIPTION:
Study design

The present study compared the effectiveness of two interventions for the treatment of PD:

1. Intermittent Anaerobic Exercise (IAE), performed as a regular and controlled systematic physical exercise of running and walking to provide Interoceptive Exposure (IE);
2. Jacobson's Progressive Muscle Relaxation method (RT). The study was designed as a prospective, two-arm, blinded, randomized, controlled clinical trial. Patients and assessors were informed that participants could receive an active pharmacological treatment or a matching placebo; however, all patients received only a placebo. The study was carried out at the Anxiety Disorders Program of the Institute of Psychiatry and the Institute of Orthopedics and Traumatology of the Faculty of Medicine of the University of São Paulo, São Paulo, Brazil.

Subjects The subjects were referred for treatment to the Anxiety Disorder Program at the emergency room (PS) of the Heart Institute (InCor). After clinical interviews of 121 suitable individuals, it was discovered that 102 met the pre-established inclusion criteria.

Participants were randomly allocated a Microsoft Excel spreadsheet to a 12-week program of IAE (n = 51) or RT (n = 51). Seventy-two patients completed the study, 38 women (52.8%) and 34 men (47.2%), aged between 21 and 51 years (mean: 33.3 ± 7.7 years). Among them, 22 (30.6%) were smokers. The mean age of onset of panic attacks was 28.3 ± 4.5 years. These groups were not significantly different in terms of sociodemographic characteristics.

Cardiovascular status assessments Initially, the subjects performed an exercise test on a medical treadmill at different speeds and inclines. As a subjective criterion, the Borg Rating of Perceived Exertion (RPE) scale was used in all tests paired with exercise intensity monitoring. However, in patients with PD, a simple assessment of subjective perception of exertion, such as the Borg RPE scale, may be insufficient to accurately capture the intensity of physical exertion. Before the test, the Physical Activity Readiness Questionnaire (PAR-Q) was used for cardiovascular risk, although the Heck test protocol presents a minimal risk of cardiac events (1/10,000-1/20,000).

Outcome evaluations The study evaluator was a trained psychiatrist with experience in using the MINI questionnaire and the rating scales used in this project. He was unaware of the patient's allocation and performed all assessments. All patients were evaluated at presentation (week -2), at baseline (week 0), and at weeks 6, 12, and 24 follow-up assessment (FU). Intervention programs were carried out weekly from week 0 to week 12.

The activities began with a short stretching session, and a warm-up, following the specificity of the exercise, of approximately 5 minutes at 55% of the individual's Maximum Heart Rate (Fcmax), previously stipulated by the exercise test (Ergospirometry).

After warming up, the patient walked for 15 minutes at 65% Fcmax. followed by a 30-second run at 85% Fcmax, returning to an active recovery of another 15 minutes of walking at 65% Fcmax, followed by another 5 minutes at 55% Fcmax, finishing with a stretch specific.

All participants had their heart rates monitored by a heart rate monitor. The time of anaerobic activity was gradually increased as a way of training this capacity and as a motivating factor for exercise.

The relaxation activities were led by a psychologist collaborating with the project. Three weekly sessions lasting 45 minutes were held. for three months. Relaxation followed criteria based on Progressive Muscle Relaxation Techniques.

The Jacobson technique can reduce or nullify the muscle tension found in anxious moments. The technique offers an easy way to identify muscles in tension and their relaxation, as most patients do not realize that the muscles are in tension.

The patient is placed in the supine position. Contract each muscle group or isolated muscle for 5 to 7 seconds and then relax for 20 to 30 seconds. The sequence is performed once, but when the region remains tense, the sequence is repeated up to 5 times. When relaxing, some verbal instructions were introduced to help with this, such as "throw away the tension", "feel calm and rested", "relax and soften your muscles" and "let the tension dissolve". The most important thing in the process was to make the patient notice the difference between muscle contraction and relaxation.

Primary outcome measure:

Changes in PD severity scores were assessed using the Panic Agoraphobia Scale (PAS), a 13-item measure of PD symptoms; Observer-rated and self-reported versions were used in the present study. The items assessed were panic attacks, agoraphobic avoidance, anticipatory anxiety, disability, functional impairment, and health concerns. The assessor was fluent in Portuguese and English and had copies of the assessed and self-reported PAS versions. The Portuguese version of the scale was translated from English by one of the authors during the scale development phase in agreement with the author.

Secondary outcome measures:

1. Frequency and intensity of panic attacks, measured through a panic attack registry;
2. Severity of general anxiety symptoms, assessed by the Hamilton Anxiety Rating Scale (HAM-A);
3. Severity of depressive symptoms, assessed by the Hamilton Rating Scale for Depression (HAM-D).

Successful response to treatment was defined as a ≥ 50% reduction from baseline scores on both Hamilton scales.

Data analysis Pearson's chi-square test was used to analyze the distribution of categorical variables. The Shapiro-Wilk test and other distribution exploration techniques were used to assess whether the continuous variables followed a normal distribution. The Mann-Whitney-U test was used to compare continuous variables between intervention groups. Two-way repeated-measures ANOVA and post-hoc analysis for pairwise comparisons with Holm's correction were used to evaluate between- and within-group differences over time.

The sample size needed for 95% power was estimated to be 36 subjects per group using G*Power software v. 3.1.9.6 (available from the University of Dusseldorf). The data were analyzed and processed using Jamovi software v. 2.2.5. A significance level of 5% was considered in all analyses.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PD with or without agoraphobia, based on the Mini International Neuropsychiatric Interview (MINI) and in accordance with the Diagnostic and Statistical Manual of mental disorders number 4 (DSM-IV) criteria;
* No undergoing medical or other treatments for at least 12 weeks.

Exclusion Criteria:

* Clinically relevant risk of cardiovascular disease (according to the Physical Activity Readiness Questionnaire - PAR-Q scale);
* Practice of regular physical exercise for ≥ 150 minutes per week;
* History or current substance abuse or dependence;
* Pregnancy;
* Breastfeeding;
* Clinically relevant suicidal ideation or previous suicide attempts.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
PD severity scores | 12 weeks of intervention
  The Panic Agoraphobia Scale scores

SECONDARY OUTCOMES:
Frequency of panic attacks | 12 weeks of intervention
  The number of panic attacks per day
Intensity of panic attacks | 12 weeks of intervention
  Intensity measured on a scale of 0 to 5, where a higher number means a greater, more severe intensity of panic attack.

OTHER OUTCOMES:
General depressive symptoms severity | 12 weeks of intervention
  Hamilton Rating Scale for Depression
General anxiety symptoms severity | 12 weeks of intervention
  Hamilton Anxiety Rating Scale

IPD SHARING:
Plan to Share IPD: No